CLINICAL TRIAL: NCT00317382
Title: Does Static Ultrasound-Preview Reduce the Incidence of Traumatic and/or Difficult Lumbar Puncture? A Randomized Control Trial
Brief Title: Does Static Ultrasound-Preview Reduce the Incidence of Difficult Lumbar Puncture?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We could not get physicians in the ED to enroll patients.
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Emergency Physician, Columbia Univeristy College of Physicians & Surgeons
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-148
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Headache; Meningitis; Subarachnoid Hemorrhage
Keywords: lumbar puncture; headache; traumatic tap
MeSH Terms: conditions — Headache; Meningitis; Subarachnoid Hemorrhage | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Ultrasound (No Intervention): Standard LP without ultrasound use
- Ultrasound Use (Experimental): Ultrasound used to assess spine and best location for lumbar puncture.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound used to visualize spine to determine best location for lumbar puncture.
  Arms: Ultrasound Use

SUMMARY:
Does the use of ultrasound facilitate a lumbar puncture by reducing the number of difficult and traumatic lumbar punctures?

DETAILED DESCRIPTION:
This is a controlled trial randomizing lumbar puncture patients to groups utilizing ultrasound to preview the bony structures of the spine versus using standard palpation technique. The goal is to determine the helpfulness of ultrasound in performing lumbar punctures (to reduce difficult and traumatic lumbar punctures) among patients whose spines cannot be easily visualized.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18
* Clinical need for lumbar puncture
* Unable to visualize spine in position for the lumbar puncture

Exclusion Criteria:

* Able to visualize the spinous processes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-12; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
3 or more needle sticks to successfully complete lumbar puncture | We collect the data immediately
Greater than 400 red blood cells in the cerebral spinal fluid | Data is obtained within 1 hour when the lab reports the results of the CSF analysis

CONTACTS AND LOCATIONS:
Overall Officials: Kaushal Shah, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St.Luke's-Roosevelt Hospital, New York, New York, United States